CLINICAL TRIAL: NCT05391815
Title: Intermediate and Long-term Efficacy of Endovascular Treatment for TASC C&D Aortoiliac Occlusive Disease: a Prospective, Multicenter, Real-world, Registry Study
Brief Title: This Study is a Prospective, Multi-center, Real World, Observational Study, Which Aims at Evaluating Intermediate and Long-term Efficacy of Endovascular Treatment for TASC C&D Aortoiliac Occlusive Disease.
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: RenJi Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Chengdu University of Traditional Chinese Medicine (Other); Xuanwu Hospital, Beijing (Other); First People's Hospital of Hangzhou (Other); Qingdao Hiser Medical Group (Other); Second Affiliated Hospital of Soochow University (Other); Liyuan Hospital of Tongji Medical College of Huazhong University of Science and Technology (Unknown); Huashan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: The ALLIANCE Study
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Aortoiliac Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, multi-center, real world, observational study, which aims at evaluating the intermediate and long-term efficacy of endovascular treatment for TASC C&D aortoiliac occlusive disease .It is estimated that 800 subjects diagnosed with TASC C&D aortoiliac occlusive disease and receive endovascular treatments will be enrolled in nine centers from April 2021 to June 2027 nation-widely. All the subjects will be under follow-up for 60 months. There is no restriction on the endovascular techniques. The primary outcomes covers freedom from TLR at 60 months.

DETAILED DESCRIPTION:
In the past decade, endovascular treatment has become the first-line treatment for iliac artery occlusion, while Aorta - bilateral femoral artery bypass surgery is preferred for more complex iliac artery occlusion. However, recently, with advances in endovascular devices and techniques, endovascular interventions have gradually replaced open surgery in many clinical problems and have shown ideal safety and efficacy.

Currently, the optimal treatment for TASC, C&D iliac artery occlusion is controversial, mostly based on limited data from single centers and few large multicenter databases or registries. In addition, the long-term efficacy of stents implantation in iliac artery disease remind unknown and might be influenced by stent type and calcification. Therefore, the purpose of this study was to evaluate the long-term efficacy and safety of endovascular treatment for TASC, C&D iliac artery occlusion in a multicenter study.

ELIGIBILITY:
Inclusion Criteria:

1. Rutherford grades 3-6.
2. Follow the follow-up arrangement.
3. Age: 18-80 years old.
4. The target lesions were in the lower abdominal aorta and/or the common iliac artery and/or the external iliac artery.
5. The stenosis degree ≥50%, or restenosis (received PTA or other adjuvant therapy, including bare or covers stents), or complete occlusion, or the presence of aortailiac artery thrombosis after PMT or CDT thrombus clearance, and then further endovascular therapy perfomred.
6. Signed informed consent.

Exclusion Criteria:

1. Known allergy to drugs used in this study, including antiplatelet or anticoagulant drugs, etc.
2. Allergy to iodine contrast agent allergy;
3. Coagulation dysfunction or hypercoagulability;
4. Breast-feeding or pregnant women;
5. Life expectancy < 24 months;
6. Body condition can not tolerate endovascular treatment;
7. Type 2B, type 3 lower limb ischemia patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The TASC C&D Aorta-iliac occlusion patients.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from clinically-driven TLR | 60 months
  CD-TLR was deﬁned as any reintervention within the target lesion(s) because of recurrent symptoms. Freedom form CD-TLR were defined as the rates of the number of patients who did not receive reintervention verse the number of patients during the follow-up period.

SECONDARY OUTCOMES:
Technical success rate | 30 days
  We defined the technical success rate as the rate of patients in whom the endovascular treatments are successfully performed.
Incidence of major adverse events. | 1month, 3 months,6 months, 12 months ,24 months
  Major adverse events include anyone of the following: all-cause mortality, Myocardial infarction, ischemic stroke, acute limb ischemia, and major amputation of a vascular etiology, and arterial thrombosis related to endovascular manipulation.
Adverser events related to insufficient lower limb blood supply. | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Major amputation, acute re-occlusion, subacute re-occlusion and chronic re-occlusion.
CD-TLR | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months
  CD-TLR was deﬁned as any reintervention within the target lesion(s) because of recurrent symptoms.
Vascular quality of life questionnaire(VascuQol) | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  The VascuQol was designed as a questionnaire containing five domains: pain (4 items), symptoms (4 items), activities (8 items), social (2 items), and emotional (7 items) to evaluate Health related quality of life (HRQL). Every item has seven response options, with scores ranging from 1 to 7. A total score is the sum of all 25 item scores divided by 25.And both the total score as well as the domain scores range from 1 (worst HRQL) to 7 (best HRQL).The lower the value, the poorer the quality of life.
Health economics evaluation | 60 months
  All the cost related to the target vessel and spent in the inpatient ward will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Indes JE, Pfaff MJ, Farrokhyar F, Brown H, Hashim P, Cheung K, Sosa JA. Clinical outcomes of 5358 patients undergoing direct open bypass or endovascular treatment for aortoiliac occlusive disease: a systematic review and meta-analysis. J Endovasc Ther. 2013 Aug;20(4):443-55. doi: 10.1583/13-4242.1. PMID 23914850
- [Background] Hajibandeh S, Hajibandeh S, Antoniou SA, Torella F, Antoniou GA. Covered vs Uncovered Stents for Aortoiliac and Femoropopliteal Arterial Disease: A Systematic Review and Meta-analysis. J Endovasc Ther. 2016 Jun;23(3):442-52. doi: 10.1177/1526602816643834. Epub 2016 Apr 20. PMID 27099281
- [Background] Stoner MC, Calligaro KD, Chaer RA, Dietzek AM, Farber A, Guzman RJ, Hamdan AD, Landry GJ, Yamaguchi DJ; Society for Vascular Surgery. Reporting standards of the Society for Vascular Surgery for endovascular treatment of chronic lower extremity peripheral artery disease. J Vasc Surg. 2016 Jul;64(1):e1-e21. doi: 10.1016/j.jvs.2016.03.420. PMID 27345516
- [Result] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Result] Tshomba Y, Melissano G, Apruzzi L, Baccellieri D, Negri G, Chiesa R. Open repair for aortic occlusive disease: indication, techniques, results, tips and tricks. J Cardiovasc Surg (Torino). 2014 Apr;55(2 Suppl 1):57-68. PMID 24796898
- [Result] Kashyap VS, Pavkov ML, Bena JF, Sarac TP, O'Hara PJ, Lyden SP, Clair DG. The management of severe aortoiliac occlusive disease: endovascular therapy rivals open reconstruction. J Vasc Surg. 2008 Dec;48(6):1451-7, 1457.e1-3. doi: 10.1016/j.jvs.2008.07.004. Epub 2008 Sep 19. PMID 18804943
- [Result] Dorigo W, Piffaretti G, Benedetto F, Tarallo A, Castelli P, Spinelli F, Fargion A, Pratesi C. A comparison between aortobifemoral bypass and aortoiliac kissing stents in patients with complex aortoiliac obstructive disease. J Vasc Surg. 2017 Jan;65(1):99-107. doi: 10.1016/j.jvs.2016.06.107. Epub 2016 Sep 12. PMID 27633164
- [Result] Rzucidlo EM, Powell RJ, Zwolak RM, Fillinger MF, Walsh DB, Schermerhorn ML, Cronenwett JL. Early results of stent-grafting to treat diffuse aortoiliac occlusive disease. J Vasc Surg. 2003 Jun;37(6):1175-80. doi: 10.1016/s0741-5214(03)00326-4. PMID 12764261
- [Result] Hans SS, DeSantis D, Siddiqui R, Khoury M. Results of endovascular therapy and aortobifemoral grafting for Transatlantic Inter-Society type C and D aortoiliac occlusive disease. Surgery. 2008 Oct;144(4):583-9; discussion 589-90. doi: 10.1016/j.surg.2008.06.021. PMID 18847642